CLINICAL TRIAL: NCT05434104
Title: Is the Naturally Occurring Prebiotic Lactoferrin an Acceptable Alternative to Antibiotic/Antifungal Tablets for Women With Bacterial Vaginosis or Thrush?
Brief Title: The LISA (Lactoferrin InStead of Antibiotics/Antifungals) Feasibility Study
Acronym: LISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St George's, University of London (Other)
Collaborators: King's College London (Other); Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021.0268
Record Dates: First submitted 2022-05-27; First posted 2022-06-27 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Bacterial Vaginosis; Candida Vaginal
Keywords: lactoferrin; prebiotic
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal | interventions — Metronidazole; Fluconazole

STUDY DESIGN:
Intervention Model Description: open label randomised feasibility study over 12 weeks with qualitative, economic and microbiological evaluations.
Who Masked: Outcomes Assessor
Masking Description: This is an open label trial and there will be no blinding to treatment allocation of the participants or researchers. However, the analysis of samples (Gram stain and microbiome analysis) will be done blind to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactoferrin intervention group (Experimental): Women will be given bovine lactoferrin 300mg vaginal pessaries to insert every evening for the first 21 days of the study [25].
  Interventions: Other: Vaginal lactoferrin
- Usual care control - standard oral antibiotics/antifungals (Active Comparator): Control women with BV will be given oral metronidazole 400mg twice daily for five days (and routine advice about avoiding alcohol). Control women with candida will be given a fluconazole 150mg capsule to take orally the same day.
  Interventions: Drug: Usual care

INTERVENTIONS:
Other: Vaginal lactoferrin — Lactoferrin vaginal pessaries to insert nightly for seven nights
  Other Names: Difesan vaginal pessaries
  Arms: Lactoferrin intervention group
Drug: Usual care — Women with bacterial vaginosis will be given oral metronidazole and women with vaginal candida will be given oral fluconazole
  Other Names: Oral metronidazole or fluconazole
  Arms: Usual care control - standard oral antibiotics/antifungals

SUMMARY:
Three-quarters of women have bacterial vaginosis (BV) or vaginal thrush/candida yeast infection at least once during their lifetime. Symptoms can include abnormal vaginal discharge, soreness, itching and an unpleasant smell. BV during pregnancy can make the baby come too early. In the UK over a million women suffer recurrent vaginal infections. These can affect their sexual relationships and quality of life, and may need repeated courses of treatment. But some women prefer not to keep taking antibiotics which can have side effects and encourage the growth of resistant superbugs.

Lactoferrin is a prebiotic protein derived from cow's milk. Women also have naturally occurring lactoferrin in their vagina where it helps to prevent infections and encourage the growth of healthy bacteria. Recent research suggests lactoferrin may be an effective treatment for BV and thrush, but this needs to be confirmed.

Aim To see if it is feasible to conduct a future trial to prove whether lactoferrin vaginal pessaries are an acceptable, effective and cost-effective alternative to antibiotic tablets for women with BV or thrush.

Methods The investigators will recruit a total of 57 women with BV and 57 with thrush from two sexual health clinics and a general practice. Women will be asked to provide self-taken vaginal samples with a cotton bud, and to complete a confidential sexual-health questionnaire. Then the women will be divided into two groups. One group will be given lactoferrin vaginal pessaries to use every night for 3-weeks. The other group will be given antibiotic/antifungal tablets. All women will be asked to provide repeat vaginal samples at home and text us about any symptoms to see if the treatment works, if the infection comes back and if they would like antibiotics. After 12-weeks all women will be invited back for a final check-up.

Outcome measures:

* Acceptability and use of vaginal lactoferrin - from questionnaires, and interviews with 15-20 women
* Recruitment and follow-up rates
* Cost of lactoferrin treatment
* The percentage of women who report their symptoms have resolved after a week
* How quickly infections clear or recur - from analysis of samples

Patient benefit:

If this study leads to a trial showing vaginal lactoferrin is an acceptable and effective alternative to antibiotics, this could help relieve symptoms, prevent antimicrobial resistance and save NHS costs.

DETAILED DESCRIPTION:
Research Question: Is it feasible to conduct a future trial to investigate if Lactoferrin is an acceptable alternative to oral antibiotics/antifungals for women with bacterial vaginosis or thrush? Background Over 200,000 women are affected by bacterial vaginosis (BV) or vaginal candida/thrush each year in England. A million women suffer recurrent infections which many find distressing. The infections may also be associated with HIV infection and adverse pregnancy outcomes. Although BV and candida can be treated with oral antibiotics/antifungals, these can have side effects and encourage the development of antimicrobial resistance, a major global health problem.

Lactoferrin is a naturally occurring prebiotic protein present in the vagina where it helps to prevent infections and normalise the vaginal microbiome. It has been used to treat refractory BV and may also be effective against candida, but more evidence is needed.

Objective To see if it is feasible to conduct a future, definitive trial in women with BV or candida to investigate if vaginal lactoferrin pessaries are as effective as oral antibiotics in resolving symptoms, preventing recurrent infection and producing a healthy lactobacilli-dominated vaginal microbiome.

Design: open label randomised feasibility study over 12 weeks with qualitative, economic and microbiological evaluations.

Setting: a sexual health clinic and a general practice

Population 114 women with genitourinary symptoms and BV (n=57) or candida (n=57) confirmed on vaginal Gram stain. After completing questionnaires and providing self-taken vaginal samples women will be randomly allocated 2:1 into intervention or control groups. All women will be followed up with repeat samples and text/online questionnaires after 1,2,3,4 and 12 weeks.

Intervention 38 women with BV and 38 women with candida will be given vaginal 300mg lactoferrin pessaries to insert nightly for 21 nights

Comparator 19 women with BV will be given metronidazole 400mg twice daily for 5-days, and 19 women with candida will be given a fluconazole 150mg capsule.

Outcomes

* Acceptability of vaginal lactoferrin - from questionnaires, and interviews
* Adherence to treatment (from participants' weekly count of remaining pessaries/tablets)
* Recruitment rate and willingness of women to be randomised
* Follow-up rate
* Acceptability of study procedures such as providing vaginal samples and responding to texts about symptoms.
* Adverse events
* Estimate of the cost of lactoferrin and the feasibility of obtaining data on healthcare use
* Percentage of participants who complete twice weekly symptom questionnaires and provide self-taken vaginal samples at home which are suitable for microbiological analyses. These findings will inform the design of a future definitive trial.

Masking

This is an open label trial and there will be no blinding to treatment allocation of the participants or researchers. However, the analysis of samples (Gram stain and microbiome analysis) will be done blind to treatment allocation [1].

Sample size calculations and analysis

We will recruit 114 women in order to achieve a final sample of 90 followed-up women at 12-weeks (30 with BV given lactoferrin, 30 with candida given lactoferrin, and 30 controls (15 with BV, 15 candida) given oral antibiotics/antifungals. This allows for 24 women (21%) either lost to follow up (12%), recruited in general practice but not BV/thrush on Gram stain (4%) or given antibiotics for an STI (3%) an unrelated reason (2%, eg dental abscess) as antibiotics may affect both symptoms and the vaginal microbiome. Sixty intervention women and 30 controls is consistent with numbers recommended by Teare et al for feasibility studies and will provide an acceptable level of precision around the study's key feasibility outcomes [32].

For example, a recruitment rate of 50% (114/228) will have a 95% confidence interval of 43.5% to 56.5%; and a follow-up rate of 80% (91 /114) will have a 95% confidence interval of 72.5% to 87.2%.

Each week the sexual health specialist investigator sees an average of six eligible women in his recurrent vaginitis clinic and the general practitioner investigator sees one or two in general practice. PPI work and our previous trials suggest ≥50% of eligible women will agree to participate [26, 27]. If we recruit an average of 3 women a week (two in clinic, one in GP) we should complete recruitment of 114 women within 38 weeks. We will allow 12 months.

Analysis of quantitative study outcomes will be descriptive. Numbers and percentages will be presented, along with 95% confidence intervals. Weekly pessary/tablet counts will be presented as mean (SD) or median (IQR) as appropriate. Numbers of adverse events and number of women with adverse events will be summarised. The flow of participants through the study will be presented in a CONSORT diagram.

Timetable (months)

1-2 set-up 3-14 recruit 114 women and randomise 2:1 to lactoferrin/standard treatment 6-19 12-week follow-up in clinic 11-20 qualitative evaluation 13-20 statistical/cost/microbiome analyses 18-23 reports/dissemination

Impact/Dissemination

Study findings will be published in high impact journals and widely publicised. If progression criteria are met, (lactoferrin is acceptable to ≥70% of women, recruitment rate≥50%, follow-up ≥70%,) this could lead to a definitive trial which confirms that treating BV/candida with lactoferrin is an acceptable, effective, safe and cost-effective alternative to antibiotics. This could benefit women by reducing their use of antibiotics, preventing recurrent infections and decreasing the spread of antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-49 years

  * Having periods (apart from women with a Mirena IUCD or polycystic ovary syndrome)
  * Ability to consent
  * Clinical diagnosis of BV or thrush confirmed on Gram stain
  * Willing to be randomised to vaginal lactoferrin pessaries or oral antibiotics/antifungals
  * Agrees to provide vaginal samples at home and post/deliver them back to the research team.
  * Agrees to avoid douching during the study (as this can flush out lactobacilli needed for a healthy microbiome).

Exclusion Criteria:

* Pregnant or breast feeding
* Currently has chlamydia, gonorrhoea or trichomonas (as treatment for these would affect the results).
* Known allergy to metronidazole or azoles
* Post-menopausal (because of diagnostic confusion between atrophic vaginitis and bacterial vaginosis)

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The acceptability of vaginal lactoferrin treatment | 4-16 weeks after recruitment
  This will be assessed from interviews with 15-20 participants
Adherence to treatment | During the first 4 weeks of the study
  This will be assessed from participants' weekly count of remaining pessaries/tablets from questionnaires at 1, 2, 3 and 4 weeks
Recruitment rate | Up to 15 months
  Investigators will record the percentage of eligible women who agree to take part
Follow-up rate | Up to 20 months
  Investigators will record the percentage of randomised women who are followed up after 12 weeks

SECONDARY OUTCOMES:
Acceptability of study procedures, and whether participants think other women would be willing to take part in a future randomised trial of lactoferrin versus oral antibiotics. | 4-16 weeks after recruitment
  Investigators will conduct telephone interviews between 4 and 16 weeks after recruitment with 15-20 participants
Adverse events such as nausea, vomiting, vaginal irritation, abdominal pain, rashes, diarrhoea | Between recruitment and 12 week follow up
  Investigators will ask about adverse events during weekly text questionnaires during the first four weeks and on the final questionnaire at 12 weeks follow up
Recurrence or persistence of infection by 12 weeks | At 12 week follow up
  Investigators will ask about symptoms of infection on the final 12 week questionnaire and assess infection status by analysis of self-taken vaginal samples
Feasibility of obtaining data on healthcare use | Last 6 months of study
  This will be assessed by comparing reported healthcare use in final 12 week questionnaires with a medical record search in 30 participants
Percentage of participants who complete twice weekly symptom questionnaires for the first four weeks after recruitment. | During the 12 weeks after recruitment
  This will be assessed from analysis of questionnaires.
Percent of self-taken samples suitable for microbiological analysis | During the 12 weeks after recruitment
  This will be assessed from microbiological analysis of self-taken vaginal samples

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Oakeshott, MD, Principal Investigator — St George's, University of London
Locations (2):
- United Kingdom (2):
  - St Thomas' NHS Trust, London
  - St George's, University of London, London

IPD SHARING:
Plan to Share IPD: No